CLINICAL TRIAL: NCT02423031
Title: Checking Out Checking In: The Development and Validation of an Electronic Screening Tool for Pediatric Psychosocial Distress
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150109; 15-M-0109
Record Dates: First submitted 2015-04-18; First posted 2015-04-22 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: Physiological Measures; Emotional Context; Pediatric; Distress Screening; Natural History
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Caregivers: caregivers of pediatric patients with cancer and other serious illnesses
- pediatric patients: pediatric patients with cancer and other serious illnesses

SUMMARY:
Background:

- Medical problems and treatments can cause stress in some people. Researchers want to learn more about how to measure distress in young people with medical illnesses. A screening tool called Checking In will be developed in order to help researchers find ways to identify concerns and stresses common to this group.

Objective:

- To create a screening tool that will help health care providers identify psychological and social distress in young people with serious illnesses.

Eligibility:

- Outpatient youth ages 8 21 who are enrolled on a research protocol at the NIH at the time of the study.

Design:

* Phase 1 participants will complete a paper-and-pencil version of Checking In. It asks about mood, pain, fatigue, peer relationships, and sleep. During this phase, participants will be asked about the wording of the questions in Checking In. They will also talk about what they thought of the questions and if they understood them.
* Phase 2 will not involve participant enrollment. During this phase the researchers will be working with technologists to develop the software for an electronic version of Checking In.
* Phase 3 participants will complete an electronic version of Checking In. Researchers will ask questions about the ease or difficulty of using an electronic screen.
* Phase 4 participants and one of their caregivers will complete an electronic version of Checking In. They will also complete other questionnaires related to mood, pain fatigue, peer relationships and sleep. They will be asked their thoughts about using Checking In. On the same day, their NIH doctor will get summary data about their questionnaire answers. The doctor will also provide feedback about the summary form.
* Researchers will compare data from Checking In with data from the other questionnaires.

DETAILED DESCRIPTION:
Objective:

The purpose of this study is to develop and implement Checking In, a brief and interactive screening measure of distress, designed to identify emotional, physical, social, practical and spiritual concerns of pediatric patients. An accompanying provider summary sheet that delineates patient report of distress, will allow providers to triage services to patients and their families, thereby enhancing patient quality of life throughout the treatment trajectory.

Objective 1: The primary objective of this protocol is to develop a brief electronic screening tool, Checking In, which would assist clinicians in assessing the presence of psychological distress in children and adolescents with cancer and other serious medical illnesses. In order to accomplish this aim, the researchers will conduct cognitive interviews with 60 pediatric patients in order to refine the questions and phrasing of items on Checking In. The results from this phase of the study of will be used to develop the electronic screen, which will be used to accomplish the remaining aims.

Objective 2: To assess the feasibility of administering Checking In to pediatric patients and their caregivers. Researchers who administer Checking In will complete a brief questionnaire rating the feasibility of administration and all barriers encountered.

Objective 3: To assess the feasibility of completing the Checking In screening tool among pediatric patients with cancer and other serious illnesses and their caregivers. This aim will be achieved by having the patients and their caregivers answer a brief questionnaire that assesses how feasible and acceptable they found Checking In to complete.

Objective 4: To establish the utility of the Checking In summary report. Providers will complete a survey evaluating the usefulness of the summary report to indicate whether: 1) the report provided useful information, 2) the information was presented in a userfriendly manner, and 3) the summary report impacted care planning for the child.

Objective 5: To assess the concurrent validity (i.e. the extent to which a test correlates with other previously validated measures of similar constructs) of Checking In as compared to validated measures of psychological symptoms (i.e. depression, anxiety, pain and fatigue) in patients with pediatric cancer, Neurofibromatosis Type 1 (NF1) or Primary Immune Deficiencies (PIDs).

Secondary Objective 1: To compare patient and caregiver ratings of Checking In in order to determine agreement rates.

-Study Population:

Outpatients, ages 8-21, enrolled in a research study either at the Pediatric Clinic or the

Primary Immune Deficiency Clinic at the NIH with a diagnosis of pediatric cancer, NF-1

LiFraumeni or PIDs will be invited to participate in this study. Additionally, outpatients

ages 8-21, receiving active cancer treatment or follow-up at Johns Hopkins, Children s

Hospital Colorado, or Levine Children s Hospital will be invited to participate.

-Design:

The initial phase of this study will consist of the researchers conducting cognitive interviews with 60 patients in order to refine the questions and phrasing of items on Checking In. Preliminary questions for Checking In were derived and modified from the PI s previous protocol on the Distress Thermometer. During this first phase, a paper and pencil version of Checking In will be used.

Results of this initial phase will be used in phase 2 to develop the electronic version of Checking In. A bid will be conducted through the NIH to hire a technology development group who will build the Checking In application. This will include the interface development, graphics, and ability for the application to generate a printout summary report. De-identified data from both phase 1 and the physician survey will be utilized to guide the application development.

During phase 3, the electronic version of Checking In will be pilot tested and assessed for feasibility. Sixty quartets, including the patient, parent/caregiver, health care provider and associated staff member will be interviewed for this phase. Patients and their parent/caregiver will be given a tablet and asked to complete Checking In. They will then be asked to complete questionnaires assessing the feasibility of the interface of the Checking In application as well as it s content. A researcher who is present to ensure that the application runs smoothly and that the interface is feasible will also complete a feasibility questionnaire evaluating the interface. Health care providers will be given the associated summary reports and asked to complete a questionnaire assessing the report content and layout as well as impact on patient care.

Once the electronic version of Checking In is finalized, researchers will begin phase 4 of the study. During phase 4, each patient will complete a brief electronic self-report distress scale, Checking In, and standardized measures of depression, anxiety, pain, fatigue, sleep disturbance, and peer relationships, as well as an evidence-based questionnaire for self-harm.

Primary caregivers will rate their child s level of distress using Checking In, as well as complete measures assessing their child s depression, anxiety, pain, fatigue, sleep disturbance, suicide risk and peer relationships

Both patients and primary caregivers will assess the feasibility of completing Checking In. Medical providers will rate the usefulness of the Checking In summary report, as well as provide a performance rating of the patient using Lansky/Karnofsky Performance status scores. Additionally, data collectors will assess the feasibility of administering Checking In in a pediatric outpatient clinic.

-Outcome Measures

Measures include Checking In; Phase 3 Feasibility Questionnaires, Phase 4 PROMIS measures of Anxiety, Depression, Fatigue, Pain Intensity, Pain Interference, Sleep Disturbance, Self Harm (evidence-based questionnaire) and Peer Relationships; and an Feasibility scale for completion of Checking In. Self- harm and suicide risk questions will only be asked to patients 10 and older.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 8 to 21 years.
* Must be enrolled in a research protocol at the NIH or receiving cancer treatment or follow-up care at Johns Hopkins, Children s Hospital Colorado, or Levine Children s Hospital and be an outpatient at time of study. The treatment protocol PI will be contacted before a patient is approached to ensure that the patient is appropriate for enrollment into this protocol.
* Must have a parent/guardian available to complete the study measures.
* Patients and caregiver must be be able to read in English and write in English (as all instruments have not been validated in other languages)

<TAB>

EXCLUSION CRITERIA:

-Patients can be excluded from this study if there is a presence of psychotic symptoms or cognitive impairment, which in the judgment of the Principal or Associate Investigator, or consulting psychiatrist would compromise the patient s ability to accurately complete the measures.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Positive score on depression, anxiety, pain and fatigue measures | Ongoing
  Positive score on depression, anxiety, pain and fatigue measures

CONTACTS AND LOCATIONS:
Overall Officials: Maryland Pao, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (4):
- United States (4):
  - Children's Hospital Colorado, Aurora, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Carolinas Medical Center Levine Children's Hospital, Charlotte, North Carolina

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-M-0109.html